CLINICAL TRIAL: NCT02276196
Title: A Phase 4, Mono-center, Randomized, Open Label, Comparator-controlled, Parallel-group, Mechanistic Intervention Trial to Assess the Effect of 8-week Treatment With the Glucagon-like Peptide-1 Receptor Agonist Lixisenatide Versus Insulin Glulisine on Renal Physiology and Biomarkers in Insulin Glargine-treated Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of LIXIsenatide on the Renal System
Acronym: ELIXIRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.H.H. Kramer, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC2014ELIX001
Record Dates: First submitted 2014-10-16; First posted 2014-10-28 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Kidney Disease; Diabetic Nephropathy; Diabetes Mellitus; Glucagon-Like Peptide 1
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus | interventions — lixisenatide; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lixisenatide (Experimental): Lixisenatide will be administered subcutaneously, once daily for 8 weeks
  Interventions: Drug: Lixisenatide
- Insulin glulisine (Active Comparator): Insulin glulisine will be administered subcutaneously, once daily for 8 weeks
  Interventions: Drug: Insulin glulisine

INTERVENTIONS:
Drug: Lixisenatide — GLP-1 receptor agonist
  Other Names: Lyxumia
  Arms: Lixisenatide
Drug: Insulin glulisine — Insulin analogue
  Other Names: Apidra
  Arms: Insulin glulisine

SUMMARY:
Based on preclinical and small-sized studies in non-diabetic individuals, incretin-based therapies, i.e. glucagon-like peptide (GLP)-1 receptor agonists and dipeptidyl peptidase-4 inhibitors, may hold promise in preventing the onset and progression of diabetic kidney disease. However, the potential renoprotective effects of these agents, that are believed to be effectuated "beyond glucose control", have not been sufficiently detailed in human diabetes.

Therefore, the present study aims to explore the mechanistic and clinical effects of GLP-1 receptor agonists on renal physiology and biomarkers in patients with type 2 diabetes.

Forty patients with insulin-treated type 2 diabetes will undergo an eight week intervention with lixisenatide or insulin glulisine in order to assess changes in the outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes (HbA1c: 6.5-10.0% or 48-86 mmol/mol)
* Stable treatment with basal insulin glargine (dose ±20%) and metformin or basal insulin glargine (dose ±20%) alone for at least 3 months
* Fasting plasma glucose <10 mmol/L or the use of >50 units of basal insulin glargine
* Females must be post-menopausal
* Caucasian
* Age: 35 - 75 years
* Body Mass Index: >25 kg/m2
* Hypertension should be under control, i.e. <140/90 mmHg, and treated with an angiotensin-converting enzyme inhibitor or angiotensin-II-receptor blocker for at least 3 months.
* Albuminuria should be treated with an angiotensin-converting enzyme inhibitor (ACE-I) or angiotensin-II-receptor blocker (ARB) for at least 3 months.

Exclusion Criteria:

* Current/chronic use of the following medication: thiazolidinediones, sulfonylurea derivatives, GLP-1 receptor agonists, dipeptidyl peptidase (DPP)-4 inhibitors, glucocorticoids, immune suppressants, antimicrobial agents, chemotherapeutics, antipsychotics, tricyclic antidepressants and monoamine oxidase inhibitors. Subjects on diuretics, will only be excluded when these drugs cannot be stopped for the duration of the study.
* Chronic use of non-steroidal anti-inflammatory drugs will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, head-ache or back ache). However, no such drugs can be taken within a time-frame of 2 weeks prior to renal-testing
* Hypoglycemia unawareness based on investigator judgment
* History of severe hypoglycemia that required emergency hospital treatment within 3 months prior to screening
* Estimated GFR <60 mL/min/1.73m2 (determined by the Modification of Diet in Renal Disease (MDRD) study equation)
* Pregnancy
* Current urinary tract infection and active nephritis
* Recent (<6 months) history of cardiovascular disease, including: acute coronary syndrome, chronic heart failure (New York Heart Association grade II-IV), stroke or transient ischemic neurologic disorder
* Complaints compatible with or established gastroparesis, neurogenic bladder and/or incomplete bladder emptying (as determined by ultrasonic bladder scan)
* Active liver disease or a 3-fold elevation of liver enzymes (aspartate aminotransferase/alanine aminotransferase) at screening
* History of or actual pancreatic disease
* History of or actual malignancy (except basal cell carcinoma)
* History of or actual severe mental disease
* Substance abuse (alcohol: defined as >4 units/day)
* Allergy to any of the agents used in the study
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate (spouse, parent, child, or sibling, whether biological or legally adopted) family of investigator site personnel directly affiliated with the study
* Inability to understand the study protocol or give informed consent

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline following 8-week treatment with a glucagon-like peptide(GLP)-1 receptor agonist versus insulin glulisine on renal hemodynamics, measured as glomerular filtration rate (GFR) / effective renal plasma flow (ERPF) | 8 weeks
  ml/min

SECONDARY OUTCOMES:
Renal damage, measured by urine biomarkers | 8 weeks
  enzyme immuno assay
Renal tubular function | 8 weeks
  e.g. percentage (%)
Blood Pressure | 8 weeks
  mmHg

OTHER OUTCOMES:
Body anthropometrics: body weight, height, body mass index, waist circumference | 8 weeks
  kilogram, meters, centimeters
Body fat content | 8 weeks
  e.g. percentage (%)
Glycemic variables | 8 weeks
  e.g. mmol/l, mmol/mol
Lipid spectrum | 8 weeks
  e.g. mmol/l
Inflammatory markers | 8 weeks
  e.g. nmol/l
Systemic hemodynamic variables | 8 weeks
  e.g. ml/min
Heart rate | 8 weeks
  beat per minute
Microvascular function | 8 weeks
  e.g. count
Arterial stiffness | 8 weeks
  e.g. augmentation index

CONTACTS AND LOCATIONS:
Locations (1):
- VU Universtiy Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Tonneijck L, Muskiet MHA, Smits MM, Hoekstra T, Kramer MHH, Danser AHJ, Diamant M, Joles JA, van Raalte DH. Postprandial renal haemodynamic effect of lixisenatide vs once-daily insulin-glulisine in patients with type 2 diabetes on insulin-glargine: An 8-week, randomised, open-label trial. Diabetes Obes Metab. 2017 Dec;19(12):1669-1680. doi: 10.1111/dom.12985. Epub 2017 Jul 25. PMID 28449402